CLINICAL TRIAL: NCT00001043
Title: A Phase I, Multicenter, Randomized Trial to Evaluate the Safety and Immunogenicity of Vaccinia-Derived MN HIV-1 Recombinant Envelope Glycoprotein (rgp160) of Human Immunodeficiency Virus at Two Different Vaccination Schedules
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Purpose: Prevention
Other Study IDs: AVEG 013B; 10560 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections; HIV Seronegativity
Keywords: Vaccines, Synthetic; Vaccinia Virus; Viral Vaccines; Smallpox Vaccine; HIV-1; HIV Envelope Protein gp160; AIDS Vaccines; HIV Seronegativity; HIV Preventive Vaccine
MeSH Terms: conditions — HIV Infections; Vaccinia

INTERVENTIONS:
Biological: gp160 Vaccine (Immuno-AG)

SUMMARY:
AMENDED 8/94: To expand the safety and immunogenicity profile of MN rgp160 vaccine (Immuno-AG) by administering a higher dose (800 mcg) at 0, 1, 6, and 12 months and 0, 2, 8 and 14 months (these two schedules were compared in VEU 013A using a dose of 200 mcg). To obtain plasma following the fourth immunization. To evaluate skin test reactivity.

ORIGINAL (replaced): To determine in healthy volunteers the safety and immunogenicity of two immunizations of MN rgp160 vaccine (Immuno-AG) in combination with a live recombinant vaccinia virus LAV HIV-1 gp160 vaccine (HIVAC-1e) versus DryVax (the standard smallpox vaccine that was used for many years) control in combination with placebo.

ORIGINAL (replaced): A gp160 vaccine derived from the MN strain, the most prevalent strain of HIV-1 in the United States, has been developed. A previous study showed that a combination vaccine strategy, consisting of priming with HIVAC-1e followed by boosting with a gp160 subunit vaccine, resulted in humoral and cellular immune responses of greater and longer duration than either vaccine alone. Thus, a live vector/subunit boost approach using the MN rgp160 vaccine merits investigation.

DETAILED DESCRIPTION:
ORIGINAL (replaced): A gp160 vaccine derived from the MN strain, the most prevalent strain of HIV-1 in the United States, has been developed. A previous study showed that a combination vaccine strategy, consisting of priming with HIVAC-1e followed by boosting with a gp160 subunit vaccine, resulted in humoral and cellular immune responses of greater and longer duration than either vaccine alone. Thus, a live vector/subunit boost approach using the MN rgp160 vaccine merits investigation.

AMENDED 8/94: Volunteers are randomized to receive 800 mcg MN rgp160 vaccine (Immuno-AG) or adjuvant control (placebo) on one of two dosing schedules. Sixteen volunteers receive candidate vaccine and four volunteers receive placebo.

ORIGINAL (replaced): Volunteers are randomized to receive either HIVAC-1e on days 0 and 56 followed by immunization with MN rgp160 vaccine on days 224 and 364, or DryVax control on days 0 and 56 followed by placebo on days 224 and 364. Ten volunteers are entered on the MN rgp160 vaccine arm and two volunteers on the placebo arm.

PER AMENDMENT 7/96: Two additional booster immunizations of 600 mcg of MN rgp 120/HIV-1 vaccine given at study months 22 and 24 to consenting St. Louis University volunteers.

ELIGIBILITY:
Inclusion Criteria

Subjects must have:

* Normal history and physical exam.
* Negative test for HIV by ELISA within 6 weeks prior to immunization.
* Negative test for HIV by Western blot.
* CD4 count >= 400 cells/mm3.
* No history of smallpox vaccination.
* Normal urine dipstick with esterase and nitrate.
* No history of immunodeficiency, chronic illness, autoimmune disease, or use of immunosuppresssive medications.

Exclusion Criteria

Co-existing Condition:

Subjects with the following conditions are excluded:

* Positive for hepatitis B surface antigen.
* Medical or psychiatric condition or occupational responsibilities that preclude compliance.
* Active syphilis (NOTE: If serology is documented to be a false positive or due to a remote (> 6 months) infection, subject is eligible).
* Active tuberculosis (NOTE: Subjects with a positive PPD and normal x-ray showing no evidence of TB and who do not require INH therapy are eligible).
* Eczema.

Household contact with persons meeting any of the following criteria:

* pregnancy, < 12 months of age, eczema, or immunodeficiency disease or use of immunosuppressive medications.

Subjects with the following prior conditions are excluded:

* History of anaphylaxis or other serious adverse reactions to vaccines.
* Eczema within the past year.
* PER 8/94 AMENDMENT: History of cancer unless surgically excised with reasonable assurance of cure.
* PER 8/94 AMENDMENT: History of serious allergic reaction requiring hospitalization or emergent medical care.

Prior Medication:

Excluded:

* Prior HIV vaccines.
* Live attenuated vaccines within the past 60 days. NOTE: Medically indicated subunit or killed vaccines (e.g., influenza, pneumococcal) do not exclude but should be administered at least 2 weeks prior to HIV immunizations.
* Experimental agents within the past 30 days.

Prior Treatment:

Excluded:

* Blood products or immunoglobulin within the past 6 months.

Higher risk behavior for HIV infection as determined by screening questionnaire, including:

* History of injection drug use within 12 months prior to study entry.
* Higher or intermediate risk sexual behavior.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Study Completion 1997-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gorse G, Study Chair
Locations (2):
- United States (2):
  - St. Louis Univ. School of Medicine AVEG, St Louis, Missouri
  - UW - Seattle AVEG, Seattle, Washington

REFERENCES:
- [Background] Gorse GJ, Corey L, Patel GB, Mandava M, Hsieh RH, Matthews TJ, Walker MC, McElrath MJ, Berman PW, Eibl MM, Belshe RB. HIV-1MN recombinant glycoprotein 160 vaccine-induced cellular and humoral immunity boosted by HIV-1MN recombinant glycoprotein 120 vaccine. National Institute of Allergy and Infectious Diseases AIDS Vaccine Evaluation Group. AIDS Res Hum Retroviruses. 1999 Jan 20;15(2):115-32. doi: 10.1089/088922299311547. PMID 10029244
- [Background] Gorse GJ, McElrath MJ, Belshe RB, Corey L, Matthews T, Eibl M, Kennedy D, Frey S, Hsieh R, Walker MC. High dose HIV-1 MN recombinant gp160 (rgp160) vaccine induces anti-v3 MN, and IgG1-4 and IgA anti-rgp160 antibodies. Int Conf AIDS. 1996 Jul 7-12;11(1):7 (abstract no MoA153)